CLINICAL TRIAL: NCT04018482
Title: Povidone Iodine vs AVEnova: A Pre-injection Disinfection Study (PAVE Study)
Acronym: PAVE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: California Retina Consultants (Other)
Responsible Party: Principal Investigator, Robert Avery, Principal Investigator, California Retina Consultants
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PAVE study
Record Dates: First submitted 2019-07-05; First posted 2019-07-12 (Actual); Last update posted 2020-03-10 (Actual); Status verified 2019-07

CONDITIONS: Age-related Macular Degeneration; Diabetic Retinopathy; Diabetic Macular Edema
Keywords: intravitreal; injection; disinfectant; comfort; Povidone Iodine; Avenova
MeSH Terms: conditions — Macular Degeneration; Diabetic Retinopathy | interventions — Povidone-Iodine; Hypochlorous Acid

STUDY DESIGN:
Intervention Model Description: A single cohort will have one eye (right) treated with Povidone Iodine (PI), and one eye (left) treated with Avenova.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Open label test arm (Experimental): Subjects will have their right eye treated with 5% Povidone Iodine per standard institutional protocol prior to receiving their intravitreal injection (2 drops of PI followed by application of 3.5% non-preserved lidocaine gel for 10 minutes, followed by 1 drop of PI for 30 seconds prior to injection). Subjects will have their left eye treated with Avenova per the same application protocol as PI prior to receiving their intravitreal injection. Prior to and following disinfecting both eyes but before the injection, a physician will gently swab the inferior conjunctival fornix (white part of each eye below the lower eye lid) with an ocular brush. Swabs will be cultured to compare bacterial counts. Subjects will be asked to complete a questionnaire regarding comfort of the disinfectant and injection procedure in general immediately following the injection and 1-2 hours post-injection.
  Interventions: Other: Povidone Iodine; Other: Hypochlorous Acid

INTERVENTIONS:
Other: Povidone Iodine — FDA-approved disinfectant for intravitreal injections
Other: Hypochlorous Acid — FDA-approved disinfectant for intravitreal injections
  Other Names: Avenova

SUMMARY:
To compare the efficacy and comfort of two FDA approved pre-injection antiseptics when used for intravitreal injections.

DETAILED DESCRIPTION:
Intravitreal injection of medicine has become the most common ocular procedure billed to Medicare. One of the main problems with this procedure is the postoperative discomfort due to the need to disinfect the eye with Povidone Iodine (PI). This disinfectant lowers the risk of endophthalmitis, but is very rough on the corneal epithelium, producing a type of corneal abrasion in many patients that is very uncomfortable in the first few days after injection. Many patients refuse the PI disinfection even though avoiding it increases the risk of endophthalmitis with the procedure. Recently another disinfectant has been FDA approved specifically for the eye to treat blepharitis and dry eye. Avenova (Av), a dilute solution of hypochlorous acid, is used several times a day for these conditions. Some practices have begun using it for PI sensitive patients before an intravitreal injection as it is FDA-approved for disinfecting peri-ocular structures. A recent in vitro study was published showing that it is superior to PI in kill times for bacteria cultured for endophthalmitis cases. Some physicians say it is superior to PI with respect to patient comfort, however, to date, there is little literature about its use for intravitreal injection. The objective of this study is to assess comfort levels between the two FDA-approved disinfection options and to compare disinfection rates between PI and Av. The hypothesis is that Av will be as effective or more effective in elimination ocular pathogens as PI and will be significantly more comfortable for patients.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be receiving same day bilateral injections of an anti-VEGF agent for any ophthalmic condition.
* Subject must be fluent in English.

Exclusion Criteria:

* Under 18 years old.
* Subjects with an allergy or adverse reaction to Povidone Iodine or Avenova.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2019-07-16 (Actual); Primary Completion 2019-08-14 (Actual); Study Completion 2019-08-14 (Actual)

PRIMARY OUTCOMES:
Comfort of Povidone Iodine vs Avenova immediately post-treatment based on an 11-point numerical scale (0-10, with 0 being no pain, and 10 being extreme pain) | Immediately following the subject's injection.
  Reported comfort levels will be collected immediately after the injection procedure. Average reported comfort levels in the Povidone Iodine group will be compared with average reported comfort levels from the Avenova group at each time point using a paired Student's T-test.
Comfort of Povidone Iodine vs Avenova 1-2 hours post treatment based on an 11-point numerical scale (0-10, with 0 being no pain, and 10 being extreme pain) | 1-2 hours post-injection.
  Reported comfort levels will be collected 1-2 hours post-injection. Average reported comfort levels in the Povidone Iodine group will be compared with average reported comfort levels from the Avenova group at each time point using a paired Student's T-test.

SECONDARY OUTCOMES:
Change in colony forming unit (CFU) growth pre- and post-treatment with Povidone Iodine or Avenova to determine if Avenova is non-inferior to Povidone Iodine for ocular disinfection. | Two time points: 30 seconds before disinfection starts (time point 0); and after the 10 minutes disinfection period and prior just prior to the injection (time point 1).
  Conjunctival swabs will be taken pre- and post-ocular disinfection and plated on Chocolate agar and blood agar. After incubating for 48 hours, average colony forming units from each agar type will be counted and the average of the ratio of [post-disinfection/pre-disinfection] will be compared between the Povisone Iodine treated eyes and the Avenova treated eyes for each agar type using a paired Student's T-Test.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Avery, MD, Principal Investigator — California Retina Consultants
Locations (1):
- California Retina Consultants, Santa Barbara, California, United States

IPD SHARING:
Plan to Share IPD: No
we do not plan to share IPD with other researchers.